CLINICAL TRIAL: NCT04208971
Title: Batch Enrollment for an Artificial Intelligence-Guided Intervention to Lower Neurologic Events in Patients With Unrecognized Atrial Fibrillation (BEAGLE)
Brief Title: Batch Enrollment for AI-Guided Intervention to Lower Neurologic Events in Unrecognized AF
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Xiaoxi Yao, Principal Investigator, Mayo Clinic
Other Study IDs: 19-012411
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BEAGLE Participants: Adult patients who have not been previously diagnosed with AF, are eligible for anticoagulation and have AI-predicted risks based on a normal sinus rhythm ECG.
  Interventions: Other: AI-enabled ECG-based Screening Tool for AF

INTERVENTIONS:
Other: AI-enabled ECG-based Screening Tool for AF — A novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based screening tool to improve atrial fibrillation diagnosis and stroke prevention.

SUMMARY:
This is a prospective study to test a novel artificial intelligence (AI)-enabled electrocardiogram (ECG)-based screening tool for improving the diagnosis of unrecognized atrial fibrillation (AF) and stroke prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Had a 10-second 12-lead ECG done at Mayo Clinic
* Men with CHA2DS2-VASc ≥2 or women with CHA2DS2-VASc ≥3

Exclusion Criteria:

* Diagnosed atrial fibrillation or atrial flutter
* Missing date of birth or sex in the electronic health record (EHR)
* A history of intracranial bleeding
* A history of end-stage kidney disease
* Have an implantable cardiac monitoring device, including a pacemaker, a defibrillator, or implanted loop recorder
* Deemed by research personnel to have limitations that would prevent them from being able to provide informed consent, use the patch, or complete interviews will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to enroll adult patients who have not been previously diagnosed with AF, are eligible for anticoagulation and have AI-predicted risks based on a normal sinus rhythm ECG.
Sampling Method: Probability Sample
Enrollment: 1225 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

PRIMARY OUTCOMES:
Diagnosis of Atrial Fibrillation as Detected by Patch Application | Three Months
  The data will be used to examine the performance of the algorithm in detecting unrecognized atrial fibrillation (e.g. positive predictive value, negative predictive value, sensitivity, specificity, and area under the curve [AUC]).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Yao, PhD, MPH, Principal Investigator — Mayo Clinic; Peter Noseworthy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Noseworthy PA, Attia ZI, Behnken EM, Giblon RE, Bews KA, Liu S, Gosse TA, Linn ZD, Deng Y, Yin J, Gersh BJ, Graff-Radford J, Rabinstein AA, Siontis KC, Friedman PA, Yao X. Artificial intelligence-guided screening for atrial fibrillation using electrocardiogram during sinus rhythm: a prospective non-randomised interventional trial. Lancet. 2022 Oct 8;400(10359):1206-1212. doi: 10.1016/S0140-6736(22)01637-3. Epub 2022 Sep 27. PMID 36179758
- [Derived] Yao X, Attia ZI, Behnken EM, Walvatne K, Giblon RE, Liu S, Siontis KC, Gersh BJ, Graff-Radford J, Rabinstein AA, Friedman PA, Noseworthy PA. Batch enrollment for an artificial intelligence-guided intervention to lower neurologic events in patients with undiagnosed atrial fibrillation: rationale and design of a digital clinical trial. Am Heart J. 2021 Sep;239:73-79. doi: 10.1016/j.ahj.2021.05.006. Epub 2021 May 24. PMID 34033803
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials